CLINICAL TRIAL: NCT00099879
Title: A Randomized, Two-Cohort Phase II Study of Two Doses of BMS-275183 Given on a Weekly Schedule in Patients With Pre-Treated Non-Small Cell Lung Cancer
Brief Title: Study of BMS-275183 in Patients With Pre-treated Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CA165-020
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BMS-275183

INTERVENTIONS:
Drug: BMS-275183

SUMMARY:
The purpose of this clinical research study is to learn if BMS-275183 can shrink or slow the growth of the cancer in subjects with non-small cell lung cancer (NSCLC). The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic pretreated NSCLC
* Measurable disease
* Adequate hematologic, hepatic and renal functions
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Inability to swallow capsules
* Recent significant cardiovascular disease
* Woman who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - Local Institution, Sacramento, California
  - Local Institution, New Haven, Connecticut
  - Local Institution, Atlanta, Georgia
  - Local Institution, Maywood, Illinois
  - Local Institution, Detroit, Michigan
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Nashville, Tennessee
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- France (3):
  - Local Institution, Besançon, Cedex
  - Local Institution, Saint-Herblain, Cedex
  - Local Institution, Belfort
- Italy (2):
  - Local Institution, Parma
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Insitution, Groningen
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- United Kingdom (2):
  - Local Institution, Shefield, Yorkshire
  - Local Institution, Manchester